CLINICAL TRIAL: NCT00804050
Title: Comparison Between Erythropoietin and Erythropoietin Associated to Differentiating Therapy With Acid 13-cis-retinoic and Dihydroxyvitamin D3 in Myelodysplastic Syndromes Without Excess of Blasts
Brief Title: Multicentric Study Comparison Between Erythropoietin and Erythropoietin Associated to Differentiating Therapy With Acid 13-cis-retinoic and Dihydroxyvitamin D3 in Myelodysplastic Syndromes Without Excess of Blasts
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties of enrollment
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Dario Ferrero, MD, University of Torino - Ospedale S Giovanni Battista
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPO2006-AISSM04; 2006-006482-16
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Erythropoietin; Acid 13-Cis-Retinoic; Dihydroxyvitamin D3; low or intermediate-1 IPSS; MDS low risk
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion A: rEPO (Experimental): rEPO for 4 mounths consequently
  Interventions: Drug: infusion A: rEPO
- Infusion B combined r-EPO (Experimental): rEPO in association with acid 13-cis-retinoic acid and Dihydroxyvitamin D3 for 4 mounths consequently
  Interventions: Drug: B Infusion rEPO combined with vitamins pills

INTERVENTIONS:
Drug: infusion A: rEPO — rEPO 40.000 unit/week for 4 mounths, then patients who have obtained an erythroid response, will continue for another 4 months with therapy rEPO. Patients who have not obtained an erythroid response, will increase the dose rEPO to 80,000 units per week for an additional 4 months.
  Arms: Infusion A: rEPO
Drug: B Infusion rEPO combined with vitamins pills — rEPO 40.000 unit/week plus acid 13 cis-retinoic (20 mg/die) plus Dihydroxyvitamin D3 (1 μg os/die), for 4 mounths. Patients who have obtained an erythroid response will continue for another 4 months with the same therapy. Patients who have not obtained an erythroid will increase the dose of rEPO to 80,000 units per week for additional 4 months.Patients also will continue with the same doses of acid 13-cis-retinoic acid and Dihydroxyvitamin D3
  Arms: Infusion B combined r-EPO

SUMMARY:
This is a prospective, randomized multicenter phase III clinical trial designed to evaluate the safety and activity of comparison between Erythropoietin and Erythropoietin Associated to Differentiating Therapy With Acid 13-Cis-Retinoic and Dihydroxyvitamin D3 in Myelodysplastic Syndromes Without Excess of Blasts

ELIGIBILITY:
Inclusion Criteria:

1. Age higher than 18;
2. Confirmed diagnosis by osseous biopsy and bone marrow cyto-morphologic counts of blast cells, of Myelodysplastic syndrome without excess of blasts: "refractary anemia", "refractary anemia with rings sideroblasts", "refractary citopenya with multilineage dysplasia", " refractary citopenya with multilineage dysplasia and rings sideroblasts" or "5q-syndrome" without excess of blasts based on WHO classification (appendix).
3. Low or intermediate-1 IPSS (appendix).
4. Hb < 11g/dl.
5. rEPO serum level < 500mU/L.
6. Women in menopause from at least one year.
7. Informed consent

Exclusion Criteria:

1. Myelodisplastic syndrome with excess of blasts (RAEB).
2. IPSS score intermediate-2 or high (appendix).
3. Forecasted allogeneic bone marrow transplant within 1 year after diagnosis(patients younger than 60 years, transfusion dependents or with serious leuko/thrombocytopenia and HLA compatible family donor).Considering the time needed to perform this procedure, the indication of a transplant from non-consanguineous donor has no contraindication to the inclusion in this protocol of the response to rEPO therapy ± differentiating therapy.
4. Renal failure with creatininemia value greater than 3 times the normal limit.
5. Chronic hepatophaty with bilirubinemia value greater than 3 times the normal limit and/or AST or ALT or ALP values greater than 5 times the normal limit.
6. Presence of second tumor or other serious pathology with life expectancy lower than one year.
7. Presence of neurologic or psychiatric pathologies that make the patient unreliable in the acquisition of drugs.
8. Allergy/intolerance known to use drugs.
9. Pregnant women.
10. Women of childbearing age or in menopause from less than one year.
11. Age < 18 years old.
12. HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
study of comparison between standard theraphy rEPO (40.000unit/week) and association therapy between rEPO (40.000unit/week)plus Acid 13-Cis-Retinoic and Dihydroxyvitamin D3 | After 8 months

SECONDARY OUTCOMES:
TO evaluate if,the patients without eritroyd response at the end of the 4° month of therapy, the increase of dose of rEPO to 80.000 U / week allows to get an increase of valued response at the end of the 8° month. | 8 months
To evaluate if there is a difference of duration in the eritroyd response with standard therapy rEPO in comparison with association therapy rEPO plus Acid 13-Cis-Retinoic and Dihydroxyvitamin D3. | 20 mounths
To evaluate the existing relationships among eritroyd response and clinical-biological parameters at baseline of anemia, subclass of MDS, silky dosing of the EPO etc. | 20 mounths
To evaluate the quality of life improvement due to therapy. | 8 mounths
To evaluate the percentage of leukemic progression. | 20 mounths

CONTACTS AND LOCATIONS:
Overall Officials: Dario Ferrero, MD, Study Director — University of Torino - Ospedale San Giovanni Battista; Alessandro Levis, MD, Study Director — Ospedale SS. Antonio, Biagio e Cesare Arrigo
Locations (18):
- Italy (18):
  - Ospedale SS. Antonio, Biagio e Cesare Arrigo, Alessandria
  - Ospedale degli Infermi, Biella
  - Spedali civili, Brescia
  - Ospedale Santo Spirito, Casale (AL)
  - Ospedale Maggiore, Chieri (TO)
  - Policlinico dell'Annunziata, Cosenza
  - Ospedale Santa Croce e Carle, Cuneo
  - Ospedale Santa Croce, Fano (PU)
  - Ospedale San Martino, Genova
  - Ospedale civile, Ivrea (TO)
  - Ospedale San Gerardo, Monza (MI)
  - Ospedale Maggiore della Carità, Novara
  - Ospedale Civile, Ovada (AL)
  - Istituto clinico Humanitas, Rozzano (MI)
  - Ospedale San Giovanni Battista Molinette, Torino
  - Ospedale Cardinale Panico, Tricase (LE)
  - Ospedale Sant'Andrea, Vercelli
  - Ospedale San Bortolo, Vicenza